CLINICAL TRIAL: NCT06679140
Title: AN INTERVENTIONAL EFFICACY AND SAFETY, PHASE 3, DOUBLE-BLIND, 2-ARM STUDY TO INVESTIGATE ORALLY ADMINISTERED IBUZATRELVIR COMPARED WITH PLACEBO IN NON-HOSPITALIZED SYMPTOMATIC ADULT AND ADOLESCENT PARTICIPANTS WITH COVID-19 WHO ARE AT HIGH RISK OF PROGRESSING TO SEVERE ILLNESS
Brief Title: A Study to Learn About a Study Medicine Called Ibuzatrelvir in Adult and Adolescent Patients With COVID-19 Who Are Not Hospitalized But Are at Risk For Severe Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C5091017; 2024-517727-39-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: COVID-19 SARS-CoV-2 Infection
Keywords: Pneumonia, Viral; Pneumonia; Respiratory Tract Infections; Infections; Virus Diseases; Coronavirus Infections; Coronaviridae Infections; Nidovirales Infections; RNA Virus Infections; Lung Diseases; Respiratory Tract Diseases; COVID-19; Viral Protease Inhibitors; Protease Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Antiviral Agents; Anti-Infective Agents; ibuzatrelvir
MeSH Terms: conditions — Pneumonia, Viral; Pneumonia; Respiratory Tract Infections; Infections; Virus Diseases; Coronavirus Infections; Coronaviridae Infections; Nidovirales Infections; RNA Virus Infections; Lung Diseases; Respiratory Tract Diseases; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind with matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ibuzatrelvir (Experimental): Ibuzatrelvir administered orally every 12 hours (twice daily) for a total of 5 days.
  Interventions: Drug: ibuzatrelvir
- placebo (Placebo Comparator): placebo administered orally every 12 hours (twice daily) for 5 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ibuzatrelvir — ibuzatrelvir tablets
  Other Names: PF-07817883
  Arms: ibuzatrelvir
Drug: placebo — placebo tablets
  Arms: placebo

SUMMARY:
The purpose of the study is to evaluate whether ibuzatrelvir is effective and safe in adults and adolescents with COVID-19 who do not need to be in the hospital but who are at high risk for progression to severe disease. Eligible participants will be randomly assigned (by chance) to receive ibuzatrelvir or matching placebo orally for 5 days. Co-administration of locally available standard of care is allowed. The total duration of the study is around 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. 12 to <18 years of age, weighing at least 40 kg, or ≥18 years of age of any weight at screening.
2. Presence of risk factors for progression to severe COVID-19 at the time of screening based on age:

   1. 12 to 49 years of age with at least two risk factors, where one must be moderate immunocompromise;
   2. 50 to 64 years of age with at least two risk factors;
   3. 65 to 74 years of age with at least one risk factor;
   4. For participants 75 years of age or older, there are no requirements related to risk factors.

   The list of risk factors includes:

   BMI ≥35 kg/m2; Current smoker; Chronic lung disease; Cardiovascular disease; Type 1 or Type 2 diabetes mellitus; Mild to moderate renal impairment; Neurodevelopmental disorders; Sickle cell disease; Moderate immunosuppression.
3. Confirmed SARS-CoV-2 infection as determined by RAT in nasal or NP specimen collected within 1 day prior to randomization. Initial onset of symptoms attributable to COVID-19 within 5 days prior to randomization and at least 1 of the specified symptoms attributable to COVID-19 present on the day of randomization. Randomization must occur no later than the 5th day, where the onset of symptoms is the first day.
4. Participants must be unable or unwilling to take nirmatrelvir/ritonavir.

Exclusion Criteria:

1. Current need or anticipated need for hospitalization within 24 hours, due to signs of severe COVID-19 illness (eg, SpO2 <94% on room air, respiratory rate >30 breaths/minute, or lung infiltrates >50%) or due to other medical conditions requiring hospitalization in the opinion of the site investigator.
2. Receiving dialysis or have known severe renal impairment [ie, eGFR consistently <30 mL/min/1.73 m2 for adults or CrCl <30 mL/min for adolescents], using the serum creatinine-based CKD-EPI formula or the Cockroft Gault, respectively.
3. Active liver disease with AST or ALT >3 ULN, Total bilirubin ≥2 × ULN (for Gilbert's syndrome, direct bilirubin >ULN is exclusionary) within the past 3 months, or liver function impairment with Class C per Child Pugh classification.
4. Suspected or confirmed concurrent active systemic infection other than COVID-19 that may interfere with the evaluation of response to the study intervention.
5. Ongoing Long COVID or Post Acute Sequelae of COVID-19 diagnosis.
6. Severely immunocompromised.
7. Any comorbidity requiring hospitalization and/or surgery within 7 days prior to study entry, or that is considered life threatening within 30 days prior to study entry, as determined by the investigator.
8. History of hypersensitivity or other contraindication to any of the components of the study interventions.
9. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
10. Current use of any prohibited concomitant medication(s).

10.Has received any other antiviral for the treatment of COVID-19, including remdesivir, nirmatrelvir/ritonavir, molnupiravir, or COVID-19 mAbs within 30 days or 5 half-lives [whichever is longer] prior to screening, or received convalescent COVID-19 plasma within 12 months.

12.Received any dose of a COVID-19 vaccine within 4 months of randomization or expected to receive one through Day 34.

13.Previous administration of an investigational product (drug or vaccine) within 30 days or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).

14.Prior participation in this clinical trial or any other clinical trial of ibuzatrelvir.

15.Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2330 (Estimated)
Dates: Start 2024-12-08 (Actual); Primary Completion 2026-12-06 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with COVID-19 related emergency department visits, all cause hospitalization and all cause mortality | Day 1 through Day 28
  The difference in proportions of patients requiring COVID 19 related emergency department visits with administration of supplemental oxygen, COVID-19 antiviral or IV treatment (eg hydration, antibiotics, or corticosteroids), all-cause hospitalization, or all-cause death through Day 28 between ibuzatrelvir and placebo, among patients who were treated ≤5 days after COVID-19 symptom onset and who were not receiving background SoC treatment for their COVID-19 infection at baseline.

SECONDARY OUTCOMES:
Time to sustained resolution of all COVID-19 targeted symptoms | Day 1 to Day 28
  The difference in median time to sustained resolution of all targeted symptoms. Symptoms will be assessed through a daily electronic diary and include sore throat, cough, fever and diarrhea, among others.
Proportion of participants with post acute COVID-19 medical events | Day 29 to Week 24
  Medical events include cardiovascular events, pulmonary events, acute kidney disease and thromboembolic events.
Proportion of participants with cardiovascular, renal and pulmonary events | Day 1 to Week 24
  Medical events include cardiovascular events, pulmonary events, acute kidney disease and thromboembolic events.
Proportion of participants with Long COVID symptoms | Day 29 to Week 24
  The difference in proportions of patients with Long COVID symptoms at Week 24. Symptoms will be assessed through a weekly electronic diary.
Changes from baseline in SARS-CoV-2 RNA levels in nasopharyngeal/nasal swabs | Day 1 through Day 34
  The viral load is measured in nasal or nasopharyngeal samples using reverse transcription polymerase chain reaction (RT-PCR)
Time to SARS-CoV-2 RNA <LLOQ | Day 1 through Day 34
  Time needed to achieve a viral load below the lower limit of quantification of the essay used to measure it.
Proportion of participants with SARS-CoV-2 RNA <LLOQ at each visit | Day 1 through Day 34
  Proportion of participants with a SARS-CoV-2 viral load below the lower limit of quantification of the essay used to measure it.
Proportion of participants with rebound in SARS-CoV-2 RNA levels in nasopharyngeal swab | Day 10 and Day 14
  Virologic rebound is defined as:
  at any follow up visit, a viral RNA level increase from End of Treatment (Day 5) of ≥ 1.0 log10 copies/mL resulting in a viral RNA level ≥3.0 log10 copies/mL.
Proportion of participants with virologic and symptomatic rebound through Day 28 | Day 10 to Day 34
  symptoms rebound is defined as: after achieving short symptom recovery (the first day of at least two consecutive diary entries where all targeted symptoms are absent), symptom rebound is the first day of at least two consecutive diary entries after Day 5 where there is any targeted symptom (regardless of severity), or when a participant is hospitalized after symptom recovery.
Proportion of participants with COVID-19-related hospitalization or all cause death through Day 28. | Day 1 to Day 28
Number of days in hospital and ICU stay in participants with hospitalization (all-cause). | Day 1 to Week 24
Number of medical visits through Week 24. | Day 1 to Week 24
  medical visits include emergency department visits, hospitalizations, visits to the general practitioner and specialist.
Proportion of participants with hospitalization (all-cause) or death (all-cause) through Week 24. | Day 1 to Week 24
Time (days) to sustained alleviation of all targeted symptoms through Day 28. | Day 1 to Day 28
  The difference in median time to sustained alleviation of all targeted symptoms. Symptoms will be assessed through a daily electronic diary and include sore throat, cough, fever and diarrhea, among others.
Proportion of participants with severe symptoms attributed to COVID-19 through Day 28. | Day 1 to Day 28
  Participants are required to record the severity of their Covid-19 symptoms over the past 24 hours daily on a 4-point scale ranging from 0 to 3, higher scores indicated more severity. The scale was reported as 0= no symptoms, 1=mild, 2=moderate and 3=severe. A participant with severe score for any targeted symptoms post-baseline is counted as severe. Percentage of participants with severe Covid-19 signs and symptoms is reported.
Duration of each targeted COVID-19 symptom. | Day 1 to Day 28
  Duration of each targeted COVID-19 symptom is defined as (First Date when the symptom achieved sustained alleviation/resolved)-(First Dose Date) + I for each participant with baseline severity of mild, moderate, or severe.
Proportion of participants with symptomatic rebound through Day 28. | Day 1 to Day 28
  Definition of symptomatic rebound: After achieving short symptom recovery (the first day of at least two consecutive diary entries where all targeted symptoms are absent), symptom rebound is the first day of at least two consecutive diary entries after Day 5 where there is any targeted symptom (regardless of severity), or when a participant is hospitalized after symptom recovery
Incidence of treatment emergent adverse events | Day 1 to Day 34
  An adverse event (AE) is any untoward medical occurrence in a participant, temporarily associated with the use of study intervention, whether or not considered related to the study intervention. Serious adverse event (SAE) is any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect; a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical events. AEs included both SAEs and all non-SAEs. An AE is considered as TEAE if the event started on or after start date of study intervention.
Incidence of SAEs and AEs leading to discontinuations. | Day 1 to Day 34

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (231):
- United States (78):
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - National Institute of Clinical Research - Bakersfield, Bakersfield, California
  - 310 Clinical Research, Inglewood, California
  - Long Beach Research Institute, Long Beach, California
  - Long Beach Clinical Trials, Long Beach, California
  - Downtown L.A. Research Center, Inc., Los Angeles, California
  - Clinica mi Salud by Focil Med, Oxnard, California
  - FOMAT Medical Research, Oxnard, California
  - Paradigm Clinical Research, LLC, Redding, California
  - Acclaim Clinical Research, San Diego, California
  - Tweedy Medical Group - Charity Health, South Gate, California
  - Breathe Clear Institute for Sinus and Allergy Relief, Torrance, California
  - Paradigm Clinical Research, LLC, Wheat Ridge, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Innovative Research of West Florida, Clearwater, Florida
  - Invictus Clinical Research Group, Coconut Creek, Florida
  - Hillcrest Medical Research LLC, DeLand, Florida
  - Hillcrest Medical Research, DeLand, Florida
  - Universal Axon Clinical Research, LLC, Doral, Florida
  - Herco Medical and Research Center Inc, Flagami, Florida
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Qway Research LLC, Hialeah, Florida
  - Sunbright Health Medical Centers, Homestead, Florida
  - Bio-Medical Research LLC, Miami, Florida
  - Kendall South Medical Center, Miami, Florida
  - Nuovida Research Center, Miami, Florida
  - Global Health Research Center, Inc., Miami Lakes, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - GCP Research, Global Clinical professionals, St. Petersburg, Florida
  - Global Health Research Center - Tampa, Tampa, Florida
  - The Hope Clinic of Emory University, Decatur, Georgia
  - Javara - Privia Medical Group Georgia - Fayetteville, Fayetteville, Georgia
  - Coastal Heritage Clinical Research, Hinesville, Georgia
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - St. Luke's Humphreys Diabetes Center, Boise, Idaho
  - St. Luke's Children's, Boise, Idaho
  - St. Luke's Elks Children's Pavilion, Boise, Idaho
  - Koch Family Medicine, Morton, Illinois
  - UL International Travel Clinic, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Centennial Medical Group, Columbia, Maryland
  - Jadestone Clinical Research, Silver Spring, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Revival Research Institute, LLC, Dearborn, Michigan
  - Henry Ford St. John Hospital, Grosse Pointe Woods, Michigan
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - McGill Family Practice, Papillion, Nebraska
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Upstate Global Health Institute, East Syracuse, New York
  - Upstate Connect Care, Syracuse, New York
  - Prime Global Research, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Remington-Davis, Inc, Columbus, Ohio
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - Zenos Clinical Research, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Southwest Mind and Body Care, Dallas, Texas
  - Memorial Hermann Hospital TMC, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - UT Physicians, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - Gulf Coast Clinical Research - Houston, Houston, Texas
  - Mercury Clinical Research - Santa Clara Family Clinic, Houston, Texas
  - The Crofoot Research Center, Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Javara - Privia Medical Group North Texas - Stephenville, Stephenville, Texas
  - Javara - Privia Medical Group Gulf Coast - Sugarland, Sugar Land, Texas
  - Mercury Clinical Research - North Houston Internal Medicine & Pediatric Clinic, Tomball, Texas
  - Alpine Research Organization, Clinton, Utah
  - Eastside Research Associates, Redmond, Washington
- Argentina (3):
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L, San Miguel de Tucumán, Tucumán Province
  - Equipo Ciencia, Buenos Aires
- Belgium (2):
  - ANIMA Research, Alken, Limburg
  - Pneumocare, Erpent
- Brazil (16):
  - Hospital Universitario Professor Edgard Santos, Salvador, Estado de Bahia
  - Infection Control, Belo Horizonte, Minas Gerais
  - School of Medicine Federal University of Minas Gerais, Belo Horizonte, Minas Gerais
  - Complexo Hospital de Clínicas da Universidade Federal do Paraná, Curitiba, Paraná
  - Centro Médico São Francisco, Curitiba, Paraná
  - Real Hospital Portugues, Recife, Pernambuco
  - Instituto Atena de Pesquisa Clinica, Natal, Rio Grande do Norte
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica - CPC/UFSM, Santa Maria, Rio Grande do Sul
  - Hospital e Maternidade Celso Pierro, Campinas, São Paulo
  - CECIP - Centro de Estudos do Interior Paulista, Jaú, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Centro de Referência e Treinamento DST/AIDS, São Paulo, São Paulo
  - Instituto Nacional de Infectologia Evandro Chagas, Rio de Janeiro
  - Instituto de Infectologia Emilio Ribas, São Paulo
- Bulgaria (13):
  - Diagnostic Consultative Center - 1 - Sevlievo EOOD, Sevlievo, Gabrovo
  - Medical Centre "Asklepiy", Dupnitsa, Kyustendil
  - SHATPD Troyan, Troyan Municipality, Lovech
  - Diagnostic Consultative Center - 1 Lom EOOD, Lom, Montana
  - MHAT Samokov, Samokov, Sofia
  - Military Medical Academy, Sofia, Sofia (stolitsa)
  - Medical Center Pulmo - 2018 EOOD, Haskovo
  - MHAT "Rahila Angelova" Pernik, Pernik
  - Diagnostic Consultative Center "Sveti Georgi" Plovdiv, Plovdiv
  - Medical Center Sveti Ivan Rilski Chudotvorets - 2010, Plovdiv
  - Ambulatory for Individual Primary Medical Care - Dr. Pavlina Petrova - Poli ET, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Diana Med 2001, Yambol
- Canada (6):
  - Vancouver Infectious Diseases Centre, Vancouver, British Columbia
  - Clinical Research of Ontario, Scarborough Village, Ontario
  - Community Care Building, Winchester, Ontario
  - Dundas Manor Nursing Home, Winchester, Ontario
  - Winchester District Memorial Hospital, Winchester, Ontario
  - Diex Recherche Quebec, Québec
- China (16):
  - The People's Hospital of Chizhou, Chizhou, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Fudan University (Xiamen Branch), Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Third Hospital of Changsha, Changsha, Hunan
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Shanghai Minhang District Central Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Ditan Hospital Capital Medical, Beijing
- Czechia (7):
  - Doktor Brno, Brno, Brno-město
  - Zdravi-fit, Protivín, Jihočeský kraj
  - MUDr. Petra První s.r.o., Radomyšl, Jihočeský kraj
  - Praktický lékař Hořiněves, Hořiněves, Královéhradecký kraj
  - Lékařský dům v Mezibranské, Prague, Praha 1
  - Ordinace Hradebni s.r.o., České Budějovice
  - ORL MUDr Pavel Navratil, Olomouc
- Denmark (5):
  - Rigshospitalet, Copenhagen, Capital Region
  - Nordsjællands Hospital - Hillerød, Hilleroed, Capital Region
  - Regionshospitalet Gødstrup, Herning, Central Jutland
  - Aalborg Universitetshospital, Syd, Aalborg, North Denmark
  - Roskilde Sygehus, Roskilde, Region Sjælland
- Finland (4):
  - FVR, Oulun rokotetutkimusklinikka, Oulu, North Ostrobothnia
  - FVR, Tampereen rokotetutkimusklinikka, Tampere, Pirkanmaa
  - FVR, Etelä-Helsingin rokotetutkimusklinikka, Helsinki, Uusimaa
  - MeVac - Meilahti Vaccine Research Center, Helsinki, Uusimaa
- Germany (7):
  - LMU Klinikum München, Munich, Bavaria
  - Praxisgemeinschaft Heimeranplatz, Munich, Bavaria
  - IKF Pneumologie Frankfurt, Clinical Research Center, Departments: Pulmonology, Endocrinology, Cardio, Frankfurt am Main, Hesse
  - Studien Rahman & Detho, Obertshausen, Hesse
  - Praxis am Ebertplatz, Cologne, North Rhine-Westphalia
  - Novopraxis Berlin GbR, Berlin
  - zibp GmbH, Berlin
- Japan (16):
  - Kamezawa Clinic, Kasugai, Aichi-ken
  - International University of Health and Welfare Narita Hospital, Narita, Chiba
  - Tashiro Endocrinology Clinic, Fukuoka, Fukuoka
  - Medical Corporation Kouhoukai Takagi Hospital, Okawa-shi, Fukuoka
  - Nishioka Hospital, Sapporo, Hokkaido
  - Terada Clinic Respiratory Medicine & General Practice, Himeji, Hyōgo
  - Koga General Hospital, Koga-shi, Ibaraki
  - Tsuchiura Beryl Clinic, Tsuchiura, Ibaraki
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - National Hospital Organization Okinawa Hospital, Ginowan, Okinawa
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Musashino Emergency Hospital, Kodaira-shi, Tokyo
  - Swing Nozaki Clinic, Musashino-shi, Tokyo
  - Yoshijima Hospital, Hiroshima
- Mexico (3):
  - Asociación Mexicana para la Investigación Clínica A.C., Pachuca, Hidalgo
  - JM Research SC, Cuernavaca, Morelos
  - Arké SMO S.A de C.V, Veracruz
- Slovakia (9):
  - IRS - Medicinska cinnost s.r.o., Vseobecna ambulancia pre dospelych, Kosice-Juh, Košice Region
  - Artromac n.o., Košice, Košice Region
  - ML MED, s.r.o., Vseobecna ambulancia pre dospelych, Moldava nad Bodvou, Košice Region
  - Plucna ambulancia Hrebenar, s.r.o., Pneumologicko-ftizeologicka ambulancia, Spišská Nová Ves, Košice Region
  - PULMO, s.r.o., Pneumologicko-ftizeologicka ambulancia, Prešov, Presov
  - MUDr. Viliam Cibik, PhD., s.r.o., Pruské, Trenčín Region
  - AMB4YOU s.r.o., Hlohovec, Trnava Region
  - VL.AK s.r.o. Vseobecna ambulancia pre dospelych, Trnava, Trnava Region
  - SALUBER SK s.r.o., Vseobecna ambulancia pre dospelych, Nové Mesto nad Váhom
- South Africa (9):
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Global Clinical Trials, Pretoria, Gauteng
  - Jongaie Research, Pretoria West, Gauteng
  - Sandton Medical Research Centre, Sandton, Gauteng
  - Dr P J Sebastian Clinical Research Centre, Chatsworth, KwaZulu-Natal
  - Synapta Clinical Research Centre, Durban, KwaZulu-Natal
  - TREAD Research, Cape Town, Western Cape
  - Langeberg Clinical Trials, Cape Town, Western Cape
  - Paarl Research Centre, Paarl, Western Cape
- South Korea (13):
  - Incheon Medical Center, Donggu, Incheon-gwangyeoksi [incheon]
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [incheon]
  - Wonju Severance Christian Hospital, Wŏnju, Kang-won-do
  - Chonnam National University Hospital, Gwangju, Kwangju-kwangyǒkshi
  - Korea University Ansan Hospital, Ansan-si, Kyǒnggi-do
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Chung-Ang University Hospital, Dongjak-gu, Seoul-teukbyeolsi [seoul]
  - Gangnam Severance Hospital, Yonsei University Health System, Gangnam-gu, Seoul-teukbyeolsi [seoul]
  - Korea University Anam Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Hallym University Kangnam Sacred Heart Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Keimyung University Dongsan Hospital, Daegu, Taegu-kwangyǒkshi
- Spain (11):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [LA Coruña]
  - Hospital Vithas Xanit Internacional, Benalmádena, Andalusia
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital Vithas Xanit Internacional, Benalmádena, Málaga
  - CHUVI- Hospital Alvaro Cunqueiro, Vigo, Pontevedra [pontevedra]
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Virgen de Valme, Seville
- Taiwan (5):
  - Far Eastern Memorial Hospital, New Taipei City, NEW Taipei
  - Tri-Service General Hospital, Taipei City, Taipei
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (8):
  - Acibadem Universitesi Atakent Hastanesi, Istanbul, İ̇stanbul
  - Ankara University Ibni Sina Hospital, Ankara
  - Hacettepe Universite Hastaneleri, Ankara
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Kocaeli Üniversitesi, Kocaeli
  - Sakarya Training and Research Hospital, Sakarya
  - Karadeniz Technical University, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091017
- See also: Pfizer Clinical Trials website — https://www.pfizerclinicaltrials.com/nct06679140-covid-19-trial